CLINICAL TRIAL: NCT04558593
Title: Surveillance of Complex Renal Cysts - The SOCRATIC Study
Acronym: SOCRATIC
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-3522
Record Dates: First submitted 2020-08-31; First posted 2020-09-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-01

CONDITIONS: Complex Renal Cyst
Keywords: renal cyst; complex cyst; Bosniak III; Bosniak IV; renal masses; active surveillance; monitoring; surgery
MeSH Terms: interventions — Watchful Waiting; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- active surveillance: 220 participants will be included in the active surveillance group. Active surveillance is close monitoring (every 6 months the first 3 years following diagnosis and annually the following years), done per standard of care Close monitoring include: abdominal imaging (ultrasound, CT or MRI), chest X-ray or CT scan and blood tests
  Interventions: Procedure: Active surveillance
- surgery: 110 participants will be included in the surgery group. Surgery is done per standard of care. The type of surgery is at the discretion of the treating physician and may include: partial resection, total resection, thermoablation.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Active surveillance — Per standard of care: Imaging and blood tests every 6 months (3 first years) and annually (following years)
  Groups: active surveillance
Procedure: Surgery — Per standard of care: partial or full resection of the kidney, imaging annually
  Groups: surgery

SUMMARY:
One third of individuals aged >60 years will be diagnosed with at least one renal cyst following abdominal imaging. These cystic lesions are categorized according to the Bosniak classification which categorizes cysts according to their degree of complexity and risk of malignancy. Growing evidence suggests that a significant proportion of Bosniak III and IV cysts are benign and that the malignant ones present low metastatic potential. Since renal surgery carries substantial morbidity (20%) and potential mortality (0.5%), active surveillance has gained attention as a potential tradeoff to surgery to overcome overtreatment. Therefore, prospective studies of long-term follow-up are needed to confirm the oncologic safety of this strategy for patients with Bosniak III/IV cysts.

This is an multicenter prospective observational longitudinal study. The main objective is to compare the 5-year follow-up cancer-specific survival between the active surveillance and the surgical groups.

DETAILED DESCRIPTION:
Background: One in three patients over 60 years old will be diagnosed with a renal cyst following abdominal imaging. Traditionally, experts have recommended that complex cystic lesions (also known as Bosniak III - IV cysts) should be surgically removed, but recent evidences suggest that many are benign or have low metastatic potential. Thus, active surveillance which involves close follow-up of a patient's condition, was proposed as a tradeoff option to surgery.

Design: Multicenter observational longitudinal prospective cohort study

Objectives: The goal of this multicenter project is to conduct a prospective study with a 5-year follow-up to confirm the oncologic outcomes of active surveillance in the management of complex cysts. The main objectives are: 1) to compare the 5-year cancer specific survival between cysts managed by surgery and active surveillance; 2) to evaluate disease progression; 3) to evaluate patient's well-being according to each management strategy; and 4) to compare the 5-year healthcare cost of both management approaches.

Study population: Patients incidentally diagnosed with a Bosniak III and/or IV cysts, who are deemed to have at least 5 years of life, and who opted to be managed by either surgery or active surveillance. (N=330)

Follow-up: Patients will DECIDE if they want to have a surgery or to be followed by active surveillance. All patients will be followed as per standard of care with either semi-annual and annual visits. Research visits will serve to assess vital status and quality of life scores (through validated questionnaires). Patients on active surveillance will also be assessed for cyst progression and might be offered invasive or systemic therapy if progression is observed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older;
* diagnosed with a Bosniak III or IV cyst (classification 2019);
* size of cystic component ≤7cm;
* cyst wall/septum nodule (obtuse margin of protrusion) <10mm (perpendicular axis) or nodular/solid component ≤2 cm in any axis;
* life expectancy >5 years (by physician's estimate);
* new diagnosis ≤ 12 months from accrual date;
* currently asymptomatic from the disease;
* deemed fit enough for surgery;
* willingness and ability to complete questionnaires in either French or English;
* able and willing to provide informed consent

Exclusion Criteria:

* history of a hereditary renal cancer syndrome;
* presence of polycystic kidney disease;
* any prior history of RCC;
* received systemic therapy for another malignancy within the 12 months prior to accrual;
* uncontrolled medical illness including infections, hypertension, arrhythmias, heart failure, or myocardial infarction/unstable angina within 6 months that would predispose to immediate surgical therapy;
* metastatic disease or evidence of vascular or nodal disease;
* unwillingness to undergo monitoring and imaging studies;
* any contra-indication(s) to contrast-enhanced imaging (estimated glomerular filtration rate <30min/mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients incidentally diagnosed with a Bosniak III or IV cysts and who opted to be managed by either surgery or active surveillance
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2029-12-20 (Estimated); Study Completion 2031-09-20 (Estimated)

PRIMARY OUTCOMES:
5-year cancer-specific survival | from the date of enrollment (defined by signed consent) to the end of follow-up (up to 5 years)
  Defined as kidney cancer survival 5 years after the enrollment

SECONDARY OUTCOMES:
5-year overall survival | from the date of enrollment (defined by signed consent) to the end of follow-up (up to 5 years)
  Defined as survival 5 years after enrollment
2-year overall survival | from the date of enrollment (defined by signed consent) up to 2 years of follow-up
  Defined as survival 2 years after enrollment
2-year cancer-specific survival | from the date of enrollment (defined by signed consent) up to 2 years of follow-up
  Defined as kidney cancer survival 2 years after the enrollment
Treatment-free survival | from the date of enrollment (defined by signed consent) up to 2 and 5 years of follow-up
  Defined as survival without treatment (in active surveillance group)
Discontinuation rate | from the date of enrollment (defined by signed consent) to the end of follow-up (up to 5 years)
  Defined as the number of people who discontinued active surveillance at the end of the study (over the total)
Tumor growth rate | if there is a progression, at the time of imaging (undefined, between 6 months and 5 years post-enrollment)
  Defined by change in volume (cm3 ) and change in maximal diameter measured over time (years). Volume will be calculated using the formula for ellipsoid volume: 0.5326 x length x width x height.
Tumor progression rate | if there is a progression, at the time of imaging (undefined, between 3 months and 5 years post-enrollment)
  Defined as the percentage of patients with tumors that have met our pre-specified progression endpoints
Time to tumor progression (Progression-free survival) | range of time from enrollment to progression (undefined, between 3 months and 5 years post-enrollment) or end of follow-up (5 years post-enrollment)
  Defined as the time from the date of enrollment to the date where an individual experienced tumor progression or censoring due to lost to follow-up or the end of follow-up period
Patient and tumor characteristics in correlation with cancer-specific death | at the baseline visit (no more than 30 days after signed consent)
  Defined as demographic (i.e. age, sex, comorbidities, medical history, etc) and tumor characteristics (i.e. tumor size, tumor complexity, etc) associated with kidney cancer deaths
Patient and tumor characteristics in correlation with disease progression | at the baseline visit (no more than 30 days after signed consent)
  Defined as demographic (i.e. age, sex, comorbidities, medical history, etc) and tumor characteristics (i.e. tumor size, tumor complexity, etc) associated with disease progression.
Perceived health change over time | range of time from enrollment to end of follow-up (maximum 5 years post-enrollment)
  Defined as the change in EQ5D-5L scores over time (enrollment to censoring due to lost of follow-up or the end of follow-up period).
Quality of life change over time | range of time from enrollment to end of follow-up (maximum 5 years post-enrollment)
  Defined as the change in short form health survey (SF-12) scores over time (enrollment to censoring due to lost of follow-up or the end of follow-up period).
Anxiety change over time | range of time from enrollment to end of follow-up (maximum 5 years post-enrollment)
  Defined as the change in Hospital Anxiety and Depression Scale (HADS) scores over time (enrollment to censoring due to lost of follow-up or the end of follow-up period).
Health cost | range of time from enrollment to end of follow-up (maximum 5 years post-enrollment)
  Defined as the total direct (patients) and indirect (healthcare system) cost associated with the management of a complex cyst according to each treatment strategy (active surveillance and surgery).

OTHER OUTCOMES:
Radiomic | On diagnostic imaging, up to 12 months prior consent form
  Predictive ability of radiomics (comparison between imaging and clinical/research data)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O Richard, MD,MSc,FRCSC, Principal Investigator — Université de Sherbrooke
Locations (18):
- Canada (17):
  - Prostate Cancer Center, Calgary, Alberta
  - Northern Alberta Urology Center, Edmonton, Alberta
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Mens Health Clinic, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - St-Joseph's Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Health Sciences Center, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Woodstock hospital, Woodstock, Ontario
  - Centre intégré de santé et de services sociaux de Chaudière-Appalaches - Hôtel-Dieu de Lévis, Lévis, Quebec
  - CHUM, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont (CISSS-EIMtl), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Centre de recherche du Centre hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - CIUSSS Mauricie-Centre-du-Québec, Trois-Rivières, Quebec
- CHU Bordeaux (URO-CCR), Bordeaux, France

IPD SHARING:
Plan to Share IPD: No